CLINICAL TRIAL: NCT02159040
Title: A 2-year, Multi-center, Phase II, Open-label, Fixed-dose, Randomized Comparative Trial of Azacitidine, With or Without Deferasirox in Patients With Higher Risk Myelodysplastic Syndromes
Brief Title: Phase II Study to Evaluate Overall Response in Patients With Higher Risk Myelodysplastic Syndromes (MDS) Treated With Azacitidine With or Without Deferasirox.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AUS47
Record Dates: First submitted 2014-05-05; First posted 2014-06-09 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: High Risk MDS
Keywords: Int-2 MDS
MeSH Terms: interventions — Azacitidine; Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azacitidine (Active Comparator): 75mg/m2 7days/28 day cycle
  Interventions: Drug: Azacitidine
- Azacitidine and Deferasirox (Experimental): azacitidine 75mg/m2 7 days/28 day cycle deferasirox 10 mg/kg/day
  Interventions: Drug: Azacitidine plus Deferasirox

INTERVENTIONS:
Drug: Azacitidine — SC or IV AZA at 75mg/m2 7 days/28 day cycle
  Arms: Azacitidine
Drug: Azacitidine plus Deferasirox — SC or IV AZA at 75mg/m2 7 days/28 day cycle DFX 10mg/kg/day
  Arms: Azacitidine and Deferasirox

SUMMARY:
The primary objective of the study is to compare the overall response rate (inclusive of complete response, partial response and hematologic improvement) per IWG 2006 criteria in patients with higher risk MDS treated with azacitidine with or without deferasirox achieved over the course of one year. Hematologic improvement must be maintained for at least 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

Male or Female, age ≥ 18 years Patients with higher risk MDS with a blast count < 20% at the time of screening IPSS Int-2 or High Risk Serum Ferritin ≥ 300 ng/mL at screening.

Sexually active women must use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal (defined as amenorrhea for at least 12 months)

Exclusion Criteria:

Patients currently receiving any therapy other than AZA for MDS (a ≥ 4 week washout period for any agent (excluding AZA) used to treat MDS prior to first dose of study treatment is required).

Patients who have received > 2 cycles of AZA or decitabine at the time of randomization. Patients who have received iron chelation therapy within 1 month of screening.

Patients who have received growth factors within 1 month of screening. Patients who have received Revlimid within 1 month of screening. Patients who have undergone hematopoietic stem cell transplant. ECOG Performance Status > 2 Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent study treatment Patients with uncontrolled systemic hypertension Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease not controlled by standard medical therapy Patients with a diagnosis of or history of clinically relevant ocular toxicity related to iron chelation Diagnosis of liver cirrhosis (either established diagnosis or diagnosis by liver biopsy or central ultrasound reading) Clinical or laboratory evidence of active Hepatitis B or Hepatitis C (HBsAg in the absence of HBsAb OR HCV Ab positive with HCV RNA positive and ALT above the normal range). History of HIV positive test result (ELISA or Western blot) Presence of a surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug Patients with an active malignancy (currently or within the past two years) with the exception of basal cell skin carcinoma or cervical carcinoma in situ or completely resected colonic polyps carcinoma in situ. History of drug or alcohol abuse within the 12 months prior to enrollment. History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative.

Patients with a known hypersensitivity to azacitidine, mannitol, or deferasirox. Calculated creatinine clearance <40mL/min Serum creatinine greater than 1.5x ULN at screening Urine protein/creatinine ratio> 1 AST or ALT greater than 3x ULN at screening Direct Bilirubin greater than 1.5x ULN at screening. Patients who received treatment with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days or are planning to receive other investigational drugs while participating in the study Patients participating in another therapeutic clinical trial Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment. Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after stopping AZA and should not father a child in this period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2015-06-26 (Actual); Study Completion 2015-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Hematology Oncology Services of Arkansas HOSA 2, Little Rock, Arkansas
  - City of Hope National Medical Center Oncology, Duarte, California
  - University of Maryland Medical Center UM Greenbaum Cancer Ctr (2), Baltimore, Maryland
  - Rochester General Hospital / Lipson Cancer Center Lipson Cancer Center, Rochester, New York
  - The Jones Clinic, Germantown, Tennessee
  - Utah Cancer Specialists IHO Corp, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ended with patient death.Only one patient in trial. No analysis will ever be done.
Period: Overall Study
Arm/Group | Azacitidine
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Per IWG 2006 Criteria
Description: ORR (inclusive of CR, PR and HI) per IWG 2006 criteria including erythroid response, platelet response and neutrophil response over the course of one year. Hematologic improvement must be maintained for at least 8 weeks in order to count as HI.
Time Frame: 1 year
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Response
Description: Time to response is defined as time from the date of the first dose of study treatment to the date of the first documented hematologic improvement.
Time Frame: up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response
Description: Duration of response is defined as time from the date of the first observed hematologic improvement to the date of the first subsequent documented disease progression or relapse per IWG 2006 criteria.
Time Frame: up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as time from the date of the first dose of study treatment to the date of the first documented disease progression or relapse per IWG 2006 criteria.
Time Frame: Up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from the date of the first dose of study treatment to the date of death from any cause.
Time Frame: up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to AML Transformation
Description: Time to AML transformation is defined as time from the date of the first dose of study treatment to the date of the first documented bone marrow blast count ≥ 20% per WHO classification 1999.
Time Frame: Up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Serum Ferritin
Description: Change in Serum Ferritin
Time Frame: up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence of Adverse Events
Description: Incidence of adverse events (AEs) overall and by severity, and serious adverse events (SAEs).
Time Frame: up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

9. Secondary Outcome: Rate of Infection
Description: Median number of infections (positive bacterial, viral or fungal culture, or infection requiring IV antimicrobial, or infection resulting in hospitalization or death) in patients treated with azacitidine alone vs. azacitidine + deferasirox
Time Frame: up to 24 months
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

10. Secondary Outcome: Prevalence of MDS/AML Related Gene Mutations
Description: Prevalence of the following mutations in the study population (TP53, EZH2, ETV6, RUNX1, ASXL1, other mutation that is present in ≥ 5% of patients)
Time Frame: Baseline
Population: Only one patient in trial. No analysis will ever be done.
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Azacitidine
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (N=1)
Death (Cardiac disorders) | 1 (1) — cardiac arrest
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (N=1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Infusion site (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No conclusion pertaining to efficacy and/or safety was drawn, only one patient was randomized to the study and their study participation was terminated prematurely due to fatal outcome of SAE.Only one patient in trial.No analysis will ever be done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.